CLINICAL TRIAL: NCT06534840
Title: Establishment and Evaluation of Moderate-severe Prediction Model of Pulmonary Complications in Liver Transplantation Patients Based on Machine Learning Algorithm
Brief Title: Evaluation of Pulmonary Complications in Liver Transplantation Patients Based on Machine Learning
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Other Study IDs: 2024HX8193
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to develop a machine learning model that predicts moderate-severe prediction model of pulmonary complications in liver transplantation patients within 14 postoperative day using a real-world, local preoperative and intraoperative electronic health records, not administrative codes.

DETAILED DESCRIPTION:
Postoperative pulmonary complications can increase the length of hospital stay and medical costs. In particular, moderate to severe pulmonary complications, which often require clinical intervention, once occur, will lead to significantly prolonged postoperative hospitalization or even cause permanent damage or death in severe cases. A number of risk-stratified cation models have been developed to identify patients at increased risk of postoperative pulmonary complications. However, these models were built by using the traditional regression analysis. However, the traditional prediction methods have the disadvantages of limited processing power of nonlinear models and outlier, and relatively single selection variables. The obtained models have poor accuracy, and the quantification degree is not enough, so it is difficult to popularize clinical application. Artificial machine learning can use it by analyzing a large number of specific features in the rich data set to identify and learn to accurately predict the diagnosis and prognosis of diseases, and surpass traditional prediction models in dealing with classification problems. The algorithms are flexible, and it is more and more widely used in clinical practice research. However, there are few reports on machine learning models predicting prognostic models related to postoperative pulmonary complications in liver transplantation patients. Therefore, we aimed to build predictive models using artificial machine learning methods to screen for their risk factors in order to provide early intervention and individualized treatment for high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years)
* Undergoing liver transplantation

Exclusion Criteria:

* Re-transplantation
* Multi-organ transplants
* Intra-operative deaths
* severe encephalopathy (West Haven criteria III or IV)
* Incomplete clinical data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent liver transplantation from January 1,2016to December 31，2019 were admitted to the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Prediction of postoperative moderate-to-severe pulmonary complications | August 2024-December 2024
  IA total of 72 variables are expected to be included, using 6 types of machine learning methods, including decision tree (DT), logistic regression (LR), random forest (, RF), support vector machine (SVM), extreme gradient lift (XGBoost), and gradient lift decision tree (GBDT) to build a moderate postoperative prediction model

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided